CLINICAL TRIAL: NCT06534515
Title: The Effect of Tomatis Auditory Stimulation in Children and Adolescent With Neurodevelopmental Disorders (TomatisOn)
Brief Title: The Effect of Tomatis Auditory Stimulation in Children and Adolescents With NDDs
Acronym: TomatisOn
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Andeea Robe, Principal Investigator, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Young researcher study
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Neurodevelopmental Disorders
Keywords: Tomatis; children; adolescents
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: This will be a two-arm, randomized controlled trial exploring whether the Tomatis training could improve the components of auditory processing in children with NDDs referred to a Romanian Child and Adolescent Psychiatric Unit. Outcomes assessment will be conducted at baseline (T1), immediately after the training (T2).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention/Treatment (Experimental): Tomatis Auditory stimulation.
  Interventions: Device: Tomatis auditory stimulation
- No intervention (No Intervention): Waitlist control.

INTERVENTIONS:
Device: Tomatis auditory stimulation — Traditional Tomatis Method Protocol
  Arms: Intervention/Treatment

SUMMARY:
The current study aims to explore the preliminary efficacy of the Tomatis method on auditory processing in children with NDDs.

DETAILED DESCRIPTION:
This will be a two-arm, randomized controlled trial exploring whether the Tomatis training could improve the components of auditory processing in children with Neurodevelopmental Disorders referred to a Romanian Child and Adolescent Psychiatric Unit. Outcomes assessment will be conducted at baseline (T1), immediately after the training (T2).

ELIGIBILITY:
Inclusion Criteria:

- neurodevelopmental disorder

Exclusion Criteria:

* intellectual disability

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Air conduction thresholds | Change from baseline AC (time 0) at immediately after the intervention (time 1)
  % Spatialization errors in air conduction
Bone conduction thresholds | Change from baseline BC(time 0) at immediately after the intervention (time 1)
  % Spatialization errors in Bone conduction

SECONDARY OUTCOMES:
Developmental Disability Children's Global Assesment Scale total score | Change from baseline DD_CGAS (time 0) at immediately after the intervention (time 1)
  Developmental Disability Children's Global Assesment Scale total score(highest score 100; superior functioning; lowest score 1: extreme impairment)

CONTACTS AND LOCATIONS:
Overall Officials: Andreea Robe, Principal Investigator — UBB
Locations (1):
- Andeea Robe, Floreşti, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerritsen, J. (2009). A Review of Research Done on Tomatis Auditory Stimulation.
- [Background] Gilmor, T. (1999). The Efficacy of the Tomatis Method for Children with Learning and Communication Disorders: A Meta-Analysis. International Journal of Listening, 13(1), 12-23. https://doi.org/10.1080/10904018.1999.10499024